CLINICAL TRIAL: NCT03860805
Title: SALpingectomy for STERilization (SALSTER); a Randomized Trial
Brief Title: SALpingectomy for STERilization (SALSTER)
Acronym: SALSTER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 316-18
Record Dates: First submitted 2018-10-30; First posted 2019-03-04 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Sterilization Tubal; Salpingectomy; Laparoscopy; Ovarian Reserve
Keywords: Sterilization Tubal; Salpingectomy; Laparoscopy; Ovarian Reserve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic tubal ligation (Active Comparator): Patients who seek for surgical permanent contraception and randomized to laparoscopic tubal ligation
  Interventions: Procedure: Laparoscopic tubal ligation
- Laparoscopic bilateral salpingectomy (Active Comparator): Patients who seek for surgical permanent contraception and randomized to laparoscopic bilateral salpingectomy
  Interventions: Procedure: Laparoscopic bilateral salpingectomy

INTERVENTIONS:
Procedure: Laparoscopic tubal ligation — Laparoscopic tubal ligation
  Arms: Laparoscopic tubal ligation
Procedure: Laparoscopic bilateral salpingectomy — Laparoscopic bilateral salpingectomy
  Arms: Laparoscopic bilateral salpingectomy

SUMMARY:
The SALSTER study is a register-based randomized clinical trial (R-RCT) that examines if laparoscopic salpingectomy instead of tubal ligation, as a contraceptive method, has no increased risk for complications and has no negative impact on ovarian function.

DETAILED DESCRIPTION:
SALSTER Study

In the last years, the management of Fallopian tubes in benign surgery has drawn a lot of attention due to rising evidence showing that some aggressive forms of ovarian cancer may originate from the distal Fallopian tubes. Concerns were raised about the implications of salpingectomy to surgical outcome and function of the ovaries. The SALSTER study attempts to evaluate the effect of salpingectomy, in regards to surgical outcomes and ovarian function, in women seeking permanent contraception with tubal ligation.

The SALSTER study is a register-based randomized clinical trial (R-RCT) that examines if laparoscopic salpingectomy instead of tubal ligation, as a contraceptive method, has no increased risk for complications and has no negative impact on ovarian function. Complications will be assessed primarily at eight weeks post-surgery according to the Clavien-Dindo classification and the existing complications questionnaires in the Swedish National Quality Register of Gynecological Surgery (GynOp). Ovarian function will be primarily assessed by determining the age of natural menopause, measured through questionnaires on bleeding pattern in GynOp every other year. Approximately 900 patients will be recruited.

In a subset of patients, the difference in Anti-Müllerian Hormone (AMH) levels from the time of surgery and 1-year after surgery will be compared between the groups. Approximately 180 patients will be recruited.

The study is expected to start in the beginning of 2019 and the first results are expected in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Planned laparoscopic sterilization
* Willing to be randomized

Exclusion Criteria:

* Women older than 49
* Not understanding the oral or written study information
* Previous malignancy involving radiation, chemotherapy or endocrine treatment affecting ovarian function

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2043-04 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications | Eight weeks post-operatively
  Complication according to the Clavien-Dindo classification or specific questions on complications in GynOp Register (Swedish National Quality Register of Gynecological Surgery). Binary data.
Age at menopause | Twenty years
  Determined from questionnaires on bleeding pattern in GynOp. Continuous data.

SECONDARY OUTCOMES:
Severe complications | Eight weeks post-operatively
  Complications according to the Clavien-Dindo classification or the specific questions on complications in GynOp. Binary data.
Operative time | At day of surgery
  In minutes. Continous data.
Perioperative blood loss | At day of surgery
  In millilitres. Continous data.
Length of hospital stay | Assessment will be done at discharge from hospital after surgery, including a period up to 8 weeks
  In Days. Continous data.
Complications according to Clavien-Dindo | One year after surgery
  Assessed according to Clavien-Dindo. Binary data.
Complications | One year after surgery
  Assessed according to the existing questions on complications in GynOp. Binary data.
Age at the start of the perimenopausal state | Up to 55 years of age
  Assessed through questionnaires in GynOp. Continous data.
Length of the perimenopausal state | Up to 55 years of age
  Assessed in GynOp. Measured in days. Continous data.
Change in menopausal symptom score | Up to 55 years of age
  Assessed with Menopause Rating Scale (MRS) in GynOp. MRS is a validated scale consisting of 11 questions, each yields a score of 1-4. Total score is reported, ranging from 4 to 44, where 4 indicates no menopausal symptoms and 44 maximum symptoms. Ordered categorical data.
Use of hormone replacement therapy at any time during follow-up | Up to 55 years of age
  Either an answer yes to question in GynOp or prescription in The Drug Prescription Register will give information on the outcome (yes/no). Binary data.
Subsequent surgery on uterus, salpinges and/or ovaries. Binary data. | At one year and up to 55 years of age
  Assessed through GynOp and through The Patient register. Both registers yield the same data (subsequent surgery yes/no). Binary data.
Pregnancy | At one year and up to 55 years of age
  Assessed in GynOp, whether pregnancy has occurred (yes/no). Binary data.
Epithelial ovarian cancer including histopathological types and grade, primary tubal and peritoneal cancer, as well as clinical stage according to International Federation of Gynecology and Obstetrics (FIGO) | 40 years
  Assessed through The Swedish Cancer Register, The Swedish Quality Register for Gynaecological Cancer, The Swedish Cause of Death Register and The Swedish Population Register. Time-to event data.
Secondary expressions of estrogen deficiency | 40 years
  Measures of fractures related to osteoporosis and cardio-vascular events will be assessed through the Patient register. Binary and time-to-event data.

OTHER OUTCOMES:
Absolute change in AMH | Measured at baseline and 1 year post-operatively
  Measured in mg/L. Continous data.

CONTACTS AND LOCATIONS:
Overall Officials: Annika Strandell, Principal Investigator — Sahlgrenska Academy
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins, E., Strandell, A., Granåsen, G., I. A. (2018). Increased risk of menopausal symptoms one year after opportunistic salpingectomy - A retrospective observational cohort study based on the Swedish National Quality Register of Gynecological Surgery. Paris: EBCOG. Retrieved from http://www.ebcog2018.org/content/detailed-program
- [Background] Dilley SE, Havrilesky LJ, Bakkum-Gamez J, Cohn DE, Michael Straughn J Jr, Caughey AB, Rodriguez MI. Cost-effectiveness of opportunistic salpingectomy for ovarian cancer prevention. Gynecol Oncol. 2017 Aug;146(2):373-379. doi: 10.1016/j.ygyno.2017.05.034. Epub 2017 Jun 1. PMID 28577884
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Falconer H, Yin L, Gronberg H, Altman D. Ovarian cancer risk after salpingectomy: a nationwide population-based study. J Natl Cancer Inst. 2015 Jan 27;107(2):dju410. doi: 10.1093/jnci/dju410. Print 2015 Feb. PMID 25628372
- [Background] Ganer Herman H, Gluck O, Keidar R, Kerner R, Kovo M, Levran D, Bar J, Sagiv R. Ovarian reserve following cesarean section with salpingectomy vs tubal ligation: a randomized trial. Am J Obstet Gynecol. 2017 Oct;217(4):472.e1-472.e6. doi: 10.1016/j.ajog.2017.04.028. Epub 2017 Apr 25. PMID 28455082
- [Background] Heinemann K, Ruebig A, Potthoff P, Schneider HP, Strelow F, Heinemann LA, Do MT. The Menopause Rating Scale (MRS) scale: a methodological review. Health Qual Life Outcomes. 2004 Sep 2;2:45. doi: 10.1186/1477-7525-2-45. PMID 15345062
- [Background] Helden JV, Weiskirchen R. Age-independent anti-Mullerian hormone (AMH) standard deviation scores to estimate ovarian function. Eur J Obstet Gynecol Reprod Biol. 2017 Jun;213:64-70. doi: 10.1016/j.ejogrb.2017.04.029. Epub 2017 Apr 18. PMID 28437631
- [Background] Kotlyar A, Gingold J, Shue S, Falcone T. The Effect of Salpingectomy on Ovarian Function. J Minim Invasive Gynecol. 2017 May-Jun;24(4):563-578. doi: 10.1016/j.jmig.2017.02.014. Epub 2017 Feb 20. PMID 28223181
- [Background] Labidi-Galy SI, Papp E, Hallberg D, Niknafs N, Adleff V, Noe M, Bhattacharya R, Novak M, Jones S, Phallen J, Hruban CA, Hirsch MS, Lin DI, Schwartz L, Maire CL, Tille JC, Bowden M, Ayhan A, Wood LD, Scharpf RB, Kurman R, Wang TL, Shih IM, Karchin R, Drapkin R, Velculescu VE. High grade serous ovarian carcinomas originate in the fallopian tube. Nat Commun. 2017 Oct 23;8(1):1093. doi: 10.1038/s41467-017-00962-1. PMID 29061967
- [Background] McKinlay SM, Brambilla DJ, Posner JG. The normal menopause transition. Maturitas. 1992 Jan;14(2):103-15. doi: 10.1016/0378-5122(92)90003-m. PMID 1565019
- [Background] Shih IeM, Kurman RJ. Ovarian tumorigenesis: a proposed model based on morphological and molecular genetic analysis. Am J Pathol. 2004 May;164(5):1511-8. doi: 10.1016/s0002-9440(10)63708-x. PMID 15111296
- [Background] Shinar S, Blecher Y, Alpern S, Many A, Ashwal E, Amikam U, Cohen A. Total bilateral salpingectomy versus partial bilateral salpingectomy for permanent sterilization during cesarean delivery. Arch Gynecol Obstet. 2017 May;295(5):1185-1189. doi: 10.1007/s00404-017-4340-x. Epub 2017 Mar 11. PMID 28285425
- [Background] Tehrani FR, Mansournia MA, Solaymani-Dodaran M, Azizi F. Age-specific serum anti-Mullerian hormone levels: estimates from a large population-based sample. Climacteric. 2014 Oct;17(5):591-7. doi: 10.3109/13697137.2014.912262. Epub 2014 Jul 9. PMID 24716733
- [Background] Trabuco EC, Moorman PG, Algeciras-Schimnich A, Weaver AL, Cliby WA. Association of Ovary-Sparing Hysterectomy With Ovarian Reserve. Obstet Gynecol. 2016 May;127(5):819-827. doi: 10.1097/AOG.0000000000001398. PMID 27054925
- [Background] Wang Y, Mang M, Wang Y, Wang L, Klein R, Kong B, Zheng W. Tubal origin of ovarian endometriosis and clear cell and endometrioid carcinoma. Am J Cancer Res. 2015 Feb 15;5(3):869-79. eCollection 2015. PMID 26045974
- [Derived] Strandell A, Magarakis L, Sundfeldt K, Palsson M, Liv P, Idahl A. Salpingectomy versus tubal occlusion in laparoscopic sterilisation (SALSTER): a national register-based randomised non-inferiority trial. Lancet Reg Health Eur. 2024 Aug 11;45:101026. doi: 10.1016/j.lanepe.2024.101026. eCollection 2024 Oct. PMID 39974774
- [Derived] Magarakis L, Idahl A, Sundfeldt K, Liv P, Palsson M, Strandell A. SALpingectomy for STERilisation (SALSTER): study protocol for a Swedish multicentre register-based randomised controlled trial. BMJ Open. 2023 Sep 4;13(9):e071246. doi: 10.1136/bmjopen-2022-071246. PMID 37666548

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03860805/SAP_002.pdf